

# TRIAL STATISTICAL ANALYSIS PLAN (MASTER)

c38787852-01

**BI Trial No.:** 1381.9

**Title:** An open-label, Phase II, platform trial evaluating safety and

efficacy of multiple BI 754091 anti-PD-1 based combination regimens in PD-(L)1 naïve and PD-(L)1 pretreated patient populations with advanced and/or metastatic solid tumours who

have had at least one line of systemic therapy

Investigational

**Product(s):** 

BI 754091 (anti-PD-1)

Responsible trial statistician(s):

Phone:

Date of statistical

20 APR 2022 SIGNED

analysis plan:

Version: Final


**Proprietary confidential information** 

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TABLE OF CONTENTS | |
|------------|------------------------------------------------|-----|
| TITLE | PAGE | 1 |
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINT(S) | 9 |
| 5.1 | PRIMARY ENDPOINT(S) | 9 |
| 5.2 | SECONDARY ENDPOINT(S) | |
| 5.2.1 | Key secondary endpoint(s) | |
| 5.2.2 | Secondary endpoint(s) | |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENT(S) | |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | SUBJECT SETS ANALYSED | |
| 6.5 | POOLING OF CENTRES | 15 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 18 |
| <b>7.</b> | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3<br>7.4 | TREATMENT COMPLIANCE | |
| 7.4.1 | PRIMARY ENDPOINT(S) Primary analysis | |
| 7.4.2 | Interim analysis | |
| 7.5 | SECONDARY ENDPOINT(S) | |
| 7.5.1 | Key secondary endpoint(s) | |
| 7.5.2 | (Other) Secondary endpoint(s) | |
| 7.7 | EXTENT OF EXPOSURE | 22. |
| <b>7.8</b> | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs. | 25 |

HISTORY TABLE......30

10.

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### LIST OF TABLES

| Table 6.1: 1 | Definition of treatment periods | 11 |
|----------------|-------------------------------------------|----|
| Table 6.2: 1 | Important protocol deviations | 12 |
| Table 6.6: 1 | Derivation rules for PFS | 16 |
| Table 6.6: 2 | Derivation rules for OS | 18 |
| Table 7.4.1: 1 | Details of confirmed BOR derivation rules | 20 |
| Table 10: 1 | History table | 30 |
| Table 6.1: 1 | Definition of treatment periods | |
| Table 6.2: 1 | Important protocol deviations | 12 |
| Table 6.6: 1 | Derivation rules for PFS | |
| Table 6.6: 2 | Derivation rules for OS | 18 |
| Table 7.4.1: 1 | Details of confirmed BOR derivation rules | 20 |
| Table 10: 1 | History table | 30 |

TSAP for BI Trial No: 1381.9 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

Include a list of all abbreviations used in the Master TSAP

| Term | Definition / description |
|---------|------------------------------------------------------------|
| AE | Adverse Event |
| BHM | Bayesian Hierarchical Model |
| CR | Complete Response |
| CTC | Common Terminology Criteria |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DBL | Database Lock |
| DC | Disease Control |
| DLT | Dose Limiting Toxicity |
| DM&SM | Boehringer Ingelheim Data Management and Statistics Manual |
| DoR | Duration of Response |
| DRA | Drug Regulatory Affairs |
| DMG | Dictionary Maintenance Group |
| ECOG | Eastern Cooperative Oncology Group |
| EMA | European Medicines Agency |
| FL | Follicular Lymphoma |
| ICH | International Conference on Harmonisation |
| IPD | Important Protocol Divations |
| iRECIST | Immune Response Evaluation Criteria in Solid Tumours |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical Quality Review Meeting |
| MTD | Maximum Tolerated Dose |
| O*C | Oracle Clinical |
| OR | Objective Response |
| OS | Overall Survival |
| PD | Progression of Disease |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetics |
| PR | Partial Response |

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|--------|-----------------------------------------------|
| PSTAT | Project Statistician |
| PT | Preferred Term |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| RECIST | Response Evaluation Criteria in Solid Tumours |
| REP | Residual Effect Period |
| RPM | Report Planning Meeting |
| SA | Statistical Analysis |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| StD | Standard Deviation |
| SMQ | Standardised MedDRA query |
| SOC | System Organ Class |
| TESS | Treatment Emergent Signs and Symptoms |
| ToC | Table of Contents |
| TMW | Trial Medical Writer |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |

#### 3. INTRODUCTION

As per ICH E9 [1], the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Master Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the Master TSAP is based on the planned analysis specification as written in Master CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, Master TSAP readers may consult the Master CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 or the latest version will be used for analyses.

R v3.5.1 and JAGS v4.3.0 or the latest versions will be used for BHM analysis.

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

In Section 2.2.2 of master CTP, Duration of immune-response (DOiR) is defined as the duration from the date of first documented iPR or iCR according to iRECIST, if applicable, as assessed by the Investigator to the date of iCPD or death among patients with iOR.

Change: Duration of iOR (DOiR), is defined as the time from first documented iCR or iPR until the earliest of disease progression (immune unconfirmed progressive disease (iUPD) that is confirmed at a later radiological assessment) or death among patients with iOR.

#### 5. ENDPOINT(S)

#### 5.1 PRIMARY ENDPOINT(S)

The primary endpoint of the trial is objective response (OR), defined as best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the Investigator.

#### 5.2 SECONDARY ENDPOINT(S)

#### 5.2.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the Master CTP.

#### 5.2.2 Secondary endpoint(s)

The secondary endpoints of the trial will include:

- Duration of response (DoR), defined as the time from first documented CR or PR (RECIST v1.1) until the earlier of disease progression or death among patients with OR.
- Disease control (DC), defined as best overall response of CR, PR, or stable disease (SD) according to RECIST v1.1 as assessed by the Investigator.
- Progression-free survival (PFS), defined as the time from first treatment until Progression of Disease (PD) or death from any cause, whichever occurs earlier.



TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT(S)

This is an open-label study. Specific dosing and treatment regimens for each of the BI 754091 combinations are described in the individual Modules.

Table 6.1: 1 Definition of treatment periods

| Analysing Treatment<br>Period | Start Date (including) | Stop Date (including) |
|---|---|---|
| Screening | Date of informed consent | Date/Time of the first<br>administration of trial<br>treatment -1 day |
| On-treatment | Date/Time of the first administration of trial treatment | Date of the last<br>administration of trial<br>treatment + REP |
| Follow up | Date of the last administration of trial treatment + REP + 1 day | Date of the last per protocol visit |

For safety analyses, adverse events (AEs) will be classified to one of the following time periods: "Screening", "On-treatment" or "Follow-up." This will be applied for all adverse events. AE reported within REP after the last trial medication will be considered on treatment. Detailed rule for assigning AEs to these time periods are listed below:

- If the date of informed consent ≤ date of AE onset or worsening of existing AE< date/time of first administration of BI 754091, then the AE is assigned to "Screening";
- If date/time of first administration of BI 754091≤ date of AE onset or worsening of existing AE ≤ date of last administration of BI 754091+ REP, then the AE is assigned to "On-treatment";
- If date of AE onset or worsening of existing AE > date of last administration of BI 754091+ REP days, then the AE is assigned to "Follow up"

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

A protocol deviation (PD) is important if it affects the rights or safety of the study subjects, or if it can potentially influence the primary outcome measurement(s) in a non-negligible way.

No per protocol set is defined for this phase II trial, but patients with IPDs will be identified and reported in the clinical trial report (CTR). Potential IPDs are defined in <u>Table 6.2: 1</u>. The final list of IPDs will be confirmed at the last report planning meeting (RPM) before data base lock (DBL).

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Important protocol deviations

| Ca<br>Co | tegory /<br>de | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| A | | Entrance criteria not met | | | |
| | A1 | Inclusion criteria not met | | | |
| | A1.1 | No confirmed diagnosis of module-specified tumor types. | Inclusion criterion (IN) 2 not met | None | Automatic |
| | A1.2 | Prior irAEs not resolved to a degree for patients moving from one module to another. | IN 3 not met | None | Automatic |
| | A1.3 | Patient < 18 years of age<br>at the time of signature of<br>ICF | IN 4 not met | None | Automatic |
| | A1.4 | ECOG score >1 | IN 5 not met | | |
| | A1.5 | Women of child-bearing potential and men able to father a child are not willing or able to use highly effective methods of birth control during trial participation and for at least 6 months after the last administration of trial medication. | IN 8 not met | None | Automatic |
| | A2 | Exclusion criteria met | | | |
| | A2.1 | Use of investigational or anti-tumour treatment within 4 weeks or within 5 half-life periods (whichever is shorter) prior to the initial administration of trial treatment. | Exclusion criterion (EX) 1 met | None | Automatic |
| | A2.2 | More than one anti-PD-<br>(L)1-based treatment<br>regimen prior to entering<br>the study. | EX 2 met | None | |
| | A2.3 | Major surgery performed<br>within 12 weeks prior to<br>first trial treatment or<br>planned within 12<br>months after screening | EX 3 met | None | Automatic |
| | A2.4 | Presence of other active invasive cancers other than the one treated in this trial within 5 years prior to screening, with the exception of appropriately treated | EX 4 met | None | Automatic |

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Category /<br>Code | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|
| | basal-cell carcinoma of<br>the skin, in situ<br>carcinoma of the uterine<br>cervix, or other local<br>tumours considered cured<br>by local treatment. | | | |
| A2.5 | Active infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at start of treatment in this trial. | EX 5 met | None | Automatic |
| A2.6 | Allogenic bone marrow or solid organ transplant. | EX 6 met | None | |
| A2.7 | Inadequate organ function or bone marrow reserve as demonstrated by the laboratory values presented in CTP Table 3.2.3: 1. | EX 7 met | None | Automatic |
| A2.8 | Any of the following cardiac criteria specified in CTP Exclusion criterion 7 | EX 8 met | None | Automatic |
| A2.9 | Known history of human immunodeficiency virus infection or an active hepatitis B or C virus infection. | EX 9 met | None | Automatic |
| A2.10 | Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy. Patients removed from previous IO therapy because of a severe immune-related adverse event (irAE). | EX 10 met | None | Automatic |
| A2.11 | Known history of severe hypersensitivity reactions to other mAbs or known hypersensitivity to the trial drugs or their excipients. | EX 11 met | None | Automatic |
| A2.12 | Known presence of<br>symptomatic central<br>nervous system (CNS)<br>metastases, unless<br>asymptomatic and off<br>corticosteroids and/or<br>anti-convulsant therapy | EX 12 met | None | |

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Ca<br>Co | tegory /<br>de | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| | | for at least 2 weeks prior | | | |
| | A2.13 | start of treatment. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment. | EX 13 met | None | Automatic |
| | A2.14 | Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial. | EX 14 met | None | Automatic |
| | A2.15 | Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes him/her an unreliable trial subject, unlikely to complete the trial, or unable to comply with the protocol procedures. | EX 15 met | None | Automatic |
| | A2.16 | Women who are pregnant, nursing, or who plan to become pregnant while in the trial and for at least 6 months after the last administration of trial medication. | EX 16 met | None | Automatic |
| | A2.17 | Men who plan to father a child while in the trial and for at least 6 months after the last administration of trial medication. | EX 17 met | None | |
| В | 7.4 | Informed consent | - 1 1 1 1 1 | | |
| | B1 | Informed consent not available/not done | Inclusion criteria 1 not met | All | Automatic |
| | B2 | Informed consent too late | Informed consent obtained later than the initiation of treatment | None | Automatic |
| C | C1.1 | Trial medication Non-compliance per | Incorrect trial medication | None | A.,,tamati 1 |
| | CI.I | protocol | dose taken or wrong dose schedule; (in fusion time, program) decision at MQRM | None | Automatic and manual |

| | itegory /<br>ode | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| | C1.2 | Discontinuation of trial medication not following the protocol | Decision at MQRM | None | Automatic and manual |
| D | | Concomitant medication | | | |
| | D1.1 | Prohibited medication use | Review concomitant medications for prohibited medication use; also refer to Section 4.2.2.1 of master the protocol or related sections in each module | None | Manual |
| E | | Study Specific | | | |
| | E1 | Incorrect study procedures performed. | Any deviation from protocol not defined above deemed important to document in study report by trial team. | TBD | Manual |

#### 6.3 SUBJECT SETS ANALYSED

#### Screened Set:

This patient set includes all patients who have signed the informed consent. The screened set will be used for patient disposition tables.

#### Treated Set (TS):

This patient set includes all patients who were documented to have received at least one dose of trial medications in at least one module. The TS is used for both efficacy analysis and safety analyses.

#### PK Analysis Set (PKS):

This patient set includes all patients in the TS with at least one valid plasma concentration. PKS will be used for all pharmacokinetic analyses



#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical analyses.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

In general missing efficacy data will not be imputed and all reasonable efforts will be taken during the trial to obtain such data. Patients with unknown vital status, missing tumour imaging data will be censored for time-to-event analyses as detailed below.

<u>Table 6.6: 1</u> describes how patients will be classified for the analysis of PFS.

Table 6.6: 1 Derivation rules for PFS

| Situation | Outcome | Date of outcome |
|---|---|---|
| No baseline radiological assessment | | |
| Patient with death on or before first planned post-baseline radiological assessment* | Event | Date of death |
| Patient without death or patient with death after first planned post-baseline radiological assessment* | Censored | Date of first treatment administration |
| Without post-baseline radiological assessme | nts | |
| Vital status is unknown or known to be alive | Censored | Date of first treatment administration |
| Death prior to or on the first planned post-<br>baseline radiological assessment* | Event | Date of death |
| Death beyond the first planned post-baseline radiological assessment* | Censored | Date of first treatment administration |
| With baseline and post-baseline radiological assessments BUT no other anti-cancer therapy | | |

| Alive and not progressed | Censored | Date of last evaluable radiological assessment |
|---|---|---|
| Progressed, no missed radiological assessment window* prior to progression | Event | Date of radiological assessment of progression |
| Progressed, but one or more consecutively missed radiological assessments window* prior to progression | Censored | Date of last evaluable radiological assessment prior to missed assessment (or first treatment administration if no post-baseline assessment prior to missed assessment) |
| Death but no progression, no missed radiological assessment window* prior to death | Event | Date of death |
| Death without progression, but one or more consecutively missed radiological assessments window* prior to death | Censored | Date of last evaluable radiological assessment prior to missed assessments |
| Initiation of subsequent anti-cancer therap | y | |
| Subsequent anti-cancer therapy started before progression or death | Censored | Date of last radiological assessment before subsequent anti-cancer therapy |
| No baseline and/or post-baseline imaging and subsequent-anti cancer therapy started prior to a death | Censored | Date of first treatment administration |

<sup>\*</sup>Refers to Table 6.7:1 in module TSAPs for first planned post-baseline radiological assessment window.

For endpoints related to OR and DC the rules defined above, where applicable, will be followed.

<u>Table 6.6: 2</u> describes how patients will be classified for the analysis of death. Patients will be censored at the date of last contact if the investigator is no longer able to contact a patient or caregiver, and vital status cannot be determined otherwise, provided that no other information indicates that the patient was near death at that point.

Table 6.6: 2 Derivation rules for OS

| Status at time of analysis | Outcome | Date of outcome |
|---|---|---|
| Death and the date of death is known | Event | Date of death |
| Death and date of death is unknown | Event | Date of last contact when the patient is known to be alive + 1 day |
| Alive | Censored | Date of last contact when the patient is known to be alive |
| Unknown | Censored | Date of last contact when the patient is known to be alive |

No other imputations will be performed on missing data although every effort will be made to obtain complete information on all AEs, with particular emphasis on potential DLTs. Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates") [2].

Missing data and outliers of PK data are handled according to [2]. PK parameters that cannot be reasonably calculated, based on the available drug concentration-time data will not be imputed.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Baseline values will be the measurements taken most recently prior to first administration of study drug in each module.

Study day will be calculated relative to the date of the first administration of study drug in each module. The day prior to first administration of study drug will be 'Day -1' and the day of first administration of study drug will be 'Day 1'; therefore 'Day 0' will not exist.

Refers to module TSAPs for specific time windows.

#### 7. PLANNED ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / Standard deviation (StD) / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to Mean, StD, Min and Max.

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated, CV (arithmetic coefficient of variation), gMean (geometric mean) and gCV (geometric coefficient of variation).

For time-to-event analysis tables the set of statistics is: number of patients [N(%)], number of patients with event [N(%)], <time to event> [months] followed by P25 (25th percentile), median, P75 (75th percentile) and number of patients censored [N(%)]. If not specified otherwise the duration as well as the time to event will be displayed in months.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

The data from each module will be analysed and reviewed together with the data from other studies in the same combination project to evaluate the safety and efficacy benefit in explored indications/patient populations. Decisions on further development will be made based on an analysis of the aggregated data for each combination via a meta-analytic approach implementing quantitative Go-NoGo rules. Results of the meta-analytic approach will be summarised as an internal research report and will be used to support the rationale and the benefit-risk assessment for future development trials, if applicable.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Descriptive statistics are planned for demographic characteristics, disease history, prior therapies, medical history, alcohol and tobacco use, baseline ECOG PS, and baseline disease assessment.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Descriptive statistics are planned for this section of the report. Concomitant diseases will be coded similarly as adverse events based on the most current Medical Dictionary for Regulatory Activities (MedDRA) version. Concomitant therapies (CTs) will be coded according to World Health Organization (WHO) Drug Dictionary. CTs will be classified according to the Anatomical Therapeutic Chemical (ATC) classification system. The third ATC level will be used to categorize CTs by therapy type. In situations where a medical product may be used for more than one equally important indication, there are often several

classification alternatives. As appropriate, patients receiving CTs with more than one possible ATC level 3 category will be counted more than once. Footnotes will clarify this possible double counting in tables.

#### 7.3 TREATMENT COMPLIANCE

Refer to module TSAPs for treatment cycles details.

#### 7.4 PRIMARY ENDPOINT(S)

#### 7.4.1 Primary analysis

For the primary endpoint objective response, will be analysed in terms of ORR, defined as the proportion of patients with best overall response of CR or PR determined according to RECIST v1.1 until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.

A BHM approach (Berry et. al., 2013) [3] will be used to derive the posterior distribution of the ORR of each patient cohort within each Module if applicable. The description of BHM approach refers to Section 7.1 in the master protocol. All calculations for the shrinkage estimator are performed using the statistical software R v3.5.1 and JAGS v4.3.0. Please refer to section 9 for more details of calculations.

Only confirmed ORR will be used for the primary analysis of the primary endpoint. Descriptive statistics regarding e.g., observed objective response rate (both confirmed and unconfirmed) for each cohort within each Module will be displayed additionally.

Confirmed best overall response will be derived according to the following derivation rules:

- If CR or PR: look at subsequent visits, if there is another CR or PR >=28 days and <= 84 days then the patient has a confirmed response. If there is not another CR or PR >=28 days and <= 84 days then the patient can be a confirmed stable disease (SD) if the CR or PR is assessed at >=35 days from the start of study treatment.
- If SD: to be confirmed SD, the measurement must have been taken at >=35 days from the start of study treatment (only one reading is necessary).
- Additional details are provided in <u>Table 7.4.1: 1</u>.

Table 7.4.1: 1 Details of confirmed BOR derivation rules

| Overall response (time point 1) | Overall response (>=28<br>and <= 84 days from<br>time point 1) | Confirmed BOR |
|---|---|---|
| CR | CR | CR |
| CR | PD | SD as long as assessed at >=35 days,, |
| | | otherwise, PD |

| CR | NE/Missing | SD as long as assessed at >=35 days, |
|-------|------------|--------------------------------------|
| | | otherwise NE |
| PR | CR | PR |
| PR | PR | PR* |
| PR | SD | SD as long as assessed at >=35 days, |
| | | otherwise PD |
| PR | PD | SD as long as assessed at >=35 days, |
| | | otherwise PD |
| PR/SD | NE/Missing | SD as long as assessed at >=35 days, |
| | | otherwise NE |
| NE | NE/Missing | NE |

<sup>\*</sup> In a scenario: PR-SD-PR, the best overall response will be derived as PR if the time window between the two PRs >=28 days and <= 84 days,.

The primary analysis will include patients who entered the trial with their initially assigned treatment, and additional analyses may be performed taking into account the patients who cross-over from different Modules if applicable.

#### 7.4.2 Interim analysis

Interim analysis will be performed when deemed necessary. Final/primary analysis for a specific treatment combination or cohort will be considered as interim analysis. A cohort or Module may be closed, if determined to be appropriate based on results on interim analyses. Note that interim analysis will not lead to any modifications within the running trial unless otherwise stated in a Module.

#### 7.5 SECONDARY ENDPOINT(S)

#### 7.5.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the CTP.

#### 7.5.2 (Other) Secondary endpoint(s)

#### **Duration of objective response**

For all patients with OR the duration of OR (DOR) will be calculated as follows:

For patients with disease progression or death or without disease progression or death (censored):

Duration of OR [days] = date of outcome – date of first assessment of OR + 1

The censoring rules for duration of OR (i.e. outcome and date of outcome) are shown in Table 6.6:1.

Kaplan-Meier estimates will be used to calculate median duration of OR for each cohort within each Module.

#### Disease control

DC will be analysed in terms of DC rate (DCR), defined as the proportion of patients with best overall response of CR, PR, SD. The same method for the analysis of primary endpoint will be used for the analysis of DC using the BHM approach. The median and 95% credible interval will be used to summarize the shrinkage estimator of DCR.

Descriptive statistics regarding e.g., observed disease control rate for each cohort within each Module will be displayed additionally.

#### **Progression-free survival**

For patients with 'event', or with "censored" as an outcome for PFS:

PFS [days] = date of outcome – date of first treatment administration + 1

The censoring rules for PFS (i.e. outcome and date of outcome) are described in <u>Table 6.6: 1</u>. The time frame for the primary assessment of PFS will be from first treatment administration until the earliest of disease progression, death or the time point of the PFS analysis.

Kaplan-Meier (KM) estimates will be used to display the distribution of PFS for each cohort on a KM curve. To support the plot estimated survival probabilities at specific time points of interest (scheduled imaging time-points) will be tabulated along with 95% confidence intervals, using Greenwood's variance estimate. In addition the survival distribution will be used to provide estimates of the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles.



#### 7.7 EXTENT OF EXPOSURE

The total number of cycles initiated and the numbers of cycle initiated will be summarized descriptively for each cohort. Refer to module TSAPs for details.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set (TS). Analysis will be performed as defined in Section 7.3.4 of the CTP.

#### 7.8.1 Adverse events

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and not on the number of AEs. The severity of AEs will be scaled according to the Common Terminology Criteria for Adverse Events (CTCAE) latest version.

AEs are collected and analysed as per the standard BI AE guideline (001-MCG-156: Handling and summarisation of adverse event data for clinical trial reports and integrated summaries) [4].

Missing and incomplete AE dates are handled as per standard BI internal guidelines (001-MCG-156 RD-01: Handling of missing and incomplete AE dates) [2].

The analyses of adverse events will be based on the concept of treatment-emergent adverse events. That means that all adverse events occurring between the first treatment administration until the end of the REP will be assigned as "on treatment".

Adverse events will be displayed by the initial dose of study medication administered on the first day of treatment.

The overall summary of adverse events will be presented.

The frequency of patients with adverse events will be summarised by treatment, primary system organ class (SOC) and preferred term (PT) for each of the following AE tables:

- All AEs by highest CTCAE grade,
- Serious AEs by highest CTCAE grade
- Investigator assessed related AEs by highest CTCAE grade
- Investigator assessed related SAEs by highest CTCAE grade
- Investigator assessed immune-related AEs by highest CTCAE grade
- Investigator assessed immune-related AEs through the whole trial
- AEs with CTCAE grade >= 3 by highest CTCAE grade
- Investigator assessed related AEs with CTCAE grade >= 3 by highest CTCAE grade
- AEs leading to treatment discontinuation by highest CTCAE grade
- AEs leading to death

Special search categories will be defined in the module TSAPs if applicable and displayed by treatment, highest CTCAE grade and PT.

Tables including only SOC without PT or the opposite may also be produced if needed.

For tables containing SOC, the sorting will be done by frequency in SOCs then frequency in PTs within SOCs. Otherwise, the tables will be sorted by frequency in PTs.

#### 7.8.2 Laboratory data

The analysis of laboratory data will be descriptive in nature and will be based on BI standards [5]. The following analyses will be performed for selected lab tests shown in table 9.2: 1:

- Descriptive statistics, including changes from baseline to worst laboratory value and from baseline to last laboratory value
- Frequency of patients with possible clinically significant abnormalities
  - o Possible clinically significance will be defined as listed in <u>Tables 9.2: 1</u>.

Analyses of descriptive statistics should use normalized lab values.

Analyses of frequencies of patients with potential clinical significance, analyses of shift, and liver function categories tables should use converted values.

Baseline for safety laboratory parameters will be the last available measurement before the start of study drug. Laboratory measurements taken between the first treatment administration until the end of the REP will be considered as on-treatment. All lab tables should be footnoted to indicate that values were excluded if they were collected after the REP.

#### Liver Function tests and potential Hy's Law

Time to initial onset of liver enzyme elevations and frequency of patients with liver enzyme elevations will be produced.

## **Boehringer Ingelheim**

c38787852-01

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

7.8.3 Vital signs

N/A

7.8.4 **ECG** 

N/A

7.8.5 **Others** 

Refer to module TSAPs for PK and biomarkers analyses.

#### 8. REFERENCES

- 1. *CPMP/ICH/363/96:* "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.
- 2. 001-MCG-156\_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON.
- 3. Berry SM, Broglio KR, Groshen S, Berry DA. Bayesian hierarchical modeling of patient subpopulations: Efficient designs of Phase II oncology clinical trial. Clinical Trials 10 (5), 720-734 (2013) [R18-2260].
- 4. 001-MCG-156: "Handling and summarization of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON.
- 5. | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON.

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.9 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

History table Table 10: 1

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial | 02-NOV-20 | | None | This is the initial TSAP with necessary information for trial conduct |
| Final | 21-FEB-21 | | None | This is the final TSAP |
| Revised | 20-APR-22 | | 6.3 | Added definition of PK Analysis Set (PKS) |
| | | | 7.4.1 | Updated confirmed best overall response derivation rule |



#### APPROVAL / SIGNATURE PAGE

Document Number: c38787852 Technical Version Number: 1.0

**Document Name:** 08-01-tsap-master-core1

**Title:** An open-label, Phase II, platform trial evaluating safety and efficacy of multiple BI 754091 anti-PD-1 based combination regimens in PD-(L)1 naïve and PD-(L)1 pretreated patient populations with advanced and/or metastatic solid tumours who have had at least one line of systemic therapy

### Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|--------------------------------|-----------|------------------------|
| Author | | 21 Apr 2022 14:49 CEST |
| Approval-Biostatistics | | 21 Apr 2022 14:54 CEST |
| Approval-Team Member Medicine | | 21 Apr 2022 15:08 CEST |
| Approval-Clinical Program | | 21 Apr 2022 16:14 CEST |
| Approval-Clinical Trial Leader | | 26 Apr 2022 15:08 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c38787852Technical Version Number:1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|